CLINICAL TRIAL: NCT06430970
Title: Prevalence Of Significant Endoscopic and Histopathologic Findings in Patients Presenting With Unexplained Iron Deficiency Anemia: A Single Center Prospective Study
Brief Title: Prevalence Of Significant Endoscopic and Histopathologic Findings in Patients Presenting With Unexplained Iron Deficiency Anemia
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Mansoura University (Other)
Responsible Party: Principal Investigator, Asmaa Gameel, Dr, Mansoura University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: MS.22.05.2001
Record Dates: First submitted 2024-05-18; First posted 2024-05-28 (Actual); Last update posted 2024-05-28 (Actual); Status verified 2024-05

CONDITIONS: Gastrointestinal Diseases
MeSH Terms: conditions — Gastrointestinal Diseases | interventions — Endoscopy

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- patients with iron deficiency anemia (Other)
  Interventions: Device: endoscopy

INTERVENTIONS:
Device: endoscopy — upper and lower endoscopy

SUMMARY:
Background In practice, however, not all anaemic patients undergo appropriate diagnostic tests for the detection of iron deficiency anemia (IDA), and a significant portion of patients with IDA do not receive endoscopic evaluations. Accordingly, this study aimed to detect the prevalence of significant endoscopic (upper and lower endoscopy) and pathological findings in patients presenting with unexplained iron deficiency anaemia.

Methods One hundred twenty-four patients with confirmed IDA with no obvious cause who visited the Internal Medicine Clinic were randomly selected. Patients with active bleeding, pregnant or lactating females, or those with contraindications to sedation were excluded. Upper and lower endoscopy were held in the endoscopy unit of Specialized Medical Hospital and tissue biopsy from significant endoscopic findings was sent for histopathological examination.

DETAILED DESCRIPTION:
Methods This is an open label prospective study conducted on one hundered twenty four patients with IDA who attended to the Endoscopy Unit, Specialized Medical hospital, Mansoura University. Patients with active bleeding, pregnant or lactating female, contraindication of sedation (uncontrolled diabetes mellitus, uncontrolled thyroid disorders, pregnancy, respiratory embarrassment) were excluded. The study protocol was approved by our ethical committee, and written consents were taken from all subjects before the procedure.

Measures All patients underwent Complete blood count (CBC) with detection of specific hematological parameters Serum ferritin, Iron and Total iron binding capacity, INR, serum albumin and bilirubin levels, ALT (Alanine Aminotransferase), AST (Aspartate aminotransferase), ESR, serum creatinine, occult blood in stool (FOBT kits ) small sample of stool collected in clean container, usually taken on consecutive days with precaution before testing include stopping non-steroidal anti-inflammatory drugs, vitamin C tablets ,raw vegetables and fruits and red meat often 48h to 72hour before test as they give false positive test (5) using immunochemical assay which detect globin chain of hemoglobin (6). All those proved with unexplained iron deficiency anemia were prepared to perform upper endoscopy and colonoscopy in later appointment.

Procedures Esophgogastroduodenoscopy and colonscopy were performed in our endoscopy unit by the same endoscopist under conscious sedation, Endoscopic examination was done by (PENTAX medical EPK-I 5000, Tokyo, Japan). We usually started with colonscopic examintion. Complete ileocolonscopy was done to all patients then esohgeogastroduoenoscopy , any macroscopic lesion was detedcted ,documented and tissue biopsy was taken and sent for histopathological examination by the same pathologist.

ELIGIBILITY:
Inclusion Criteria:

* • Sex: both

  * Age: from 18 to 70 years
  * Cases confirmed iron deciency anemia with no obvious cause.
  * Significant UGI pathology includes Barrett's esophagus, esophagitis (LA class ≥ C), esophagogastric varices, peptic ulcer disease, duodenal ulcer, angioectasia , and cancer (Wuerth BA and Rockey DC,2018).
  * Significant LGI pathology includes adenomatous polyps >1cm, angioectasias, rectal ulcer, IBS , colon polyps and cancer. ( Ghassemi KA and Jensen DM,2013).

Exclusion Criteria:

* Patients with active bleeding, pregnant or lactating female, contraindication of sedation (uncontrolled diabetes mellitus, uncontrolled thyroid disorders, pregnancy, respiratory embarrassment) were excluded.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 124 (Estimated)
Dates: Start 2023-01-01 (Actual); Primary Completion 2025-01-01 (Estimated); Study Completion 2025-01-01 (Estimated)

PRIMARY OUTCOMES:
diagnosis of the cause of anemia | two years

CONTACTS AND LOCATIONS:
Locations (1):
- Mansoura University, Al Mansurah, Dakhlia, Egypt

IPD SHARING:
Plan to Share IPD: Undecided